CLINICAL TRIAL: NCT00245934
Title: Observational Study With Enbrel in Patients With Rheumatoid Arthritis
Brief Title: Study Evaluating Enbrel in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101354
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Enbrel

SUMMARY:
The purpose of this study is to investigate the incidence of adverse events for patients with rheumatoid arthritis treated with Enbrel under usual care settings. In addition, differences in injection site reactions based on whether health care professionals or patients administer Enbrel will be assessed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Proven diagnosis of rheumatoid arthritis

Exclusion Criteria:

* Contraindications according to Summary of Product Characteristic (SmPC)of Enbrel® the following points will prevent or restrict participation:

  * Patients who suffer from hypersensitivity to the active substance Etanercept or to any of the excipients of Enbrel®
  * Treatment with Enbrel® should not be initiated in patients with active infections including chronic or localized infections
  * Patients with sepsis or risk of sepsis should not be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2003-06; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com